CLINICAL TRIAL: NCT04531436
Title: Testing a Brief Mindful Eating Program: Feasibility and Proof of Concept
Brief Title: Testing a Brief Mindful Eating Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Barbel Knauper, James McGill Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46-0617
Record Dates: First submitted 2020-08-11; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Overeating; Overweight; Obesity
Keywords: Mindful eating; Overweight; Obesity; Intuitive eating; Overeating; Self-compassion
MeSH Terms: conditions — Hyperphagia; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Pilot feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Brief mindful eating intervention
  Interventions: Other: Brief mindful eating intervention

INTERVENTIONS:
Other: Brief mindful eating intervention — Over the 9-week intervention, participants will be introduced to various mindful eating and intuitive eating practices which are aimed at reducing overeating and facilitating weight loss. Each session will focus on one simple, evidence-based message, aimed at modifying a current weight-relevant eating behavior of the patient. The intervention will focus on two key elements: (1) the mindful awareness of body cues (intuitive eating) and (2) the mindful awareness of external cues (mindful eating).

SUMMARY:
This project evaluated the effects of a brief manualized mindful eating intervention as a treatment for overeating with individuals with overweight and obesity.

DETAILED DESCRIPTION:
Overeating leads to overweight and obesity. Effective eating regulation largely depends on an individual's responsiveness to internal cues of physiological hunger and satiety; this phenomenon is known as interoceptive awareness and has been shown to be lower in individuals with overweight or obesity. Mindfulness training may improve interoceptive awareness and thus may facilitate more effective regulation of eating through increased sensitivity to cues of hunger and fullness. Mindful eating programs have been shown to increase interoceptive awareness of hunger and satiety cues and decrease weight in individuals with obesity. Although these programs are effective, they involve lengthy group sessions, require extensively trained staff, and are not widely available outside of clinical research. Thus, the reach and impact of these programs are limited.

The present study developed and tested a brief mindful eating intervention inspired by Kristeller & Wolever's (2010) Mindfulness-Based Eating Awareness Training program to increase interoceptive awareness in individuals with overweight and obesity as a means to increase mindful and intuitive eating, reduce overeating and facilitate weight loss. The program consisted of 9 weekly 10-15 minute sessions structured around one simple evidence-based mindful eating exercise, and was delivered to adult (ages 18-67) employees from a Canadian university.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 25 to 45 kg/m2 (overweight/obese)
* Willingness to commit to program and complete various assessment measures

Exclusion Criteria:

* Having been pregnant in the past six months or planning on becoming pregnant in the next year
* Undergoing treatment for cancer
* Using medications that affect body weight or appetite
* Being diagnosed with bulimia nervosa, binge-eating disorder, major depressive disorder, or another severe psychiatric disease (including dementia)

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Change in overeating | Baseline, week 9, and 24-week follow-up
  As measured by the Overeating Questionnaire. Scores can range from 0 to 40, with higher scores indicating a greater tendency to overeat

SECONDARY OUTCOMES:
Change in body weight | Baseline, week 9, and 24-week follow-up
  Change in body weight (lbs)

OTHER OUTCOMES:
Change in mindful eating | Baseline, week 7, 24-week follow-up
  As measured by the Mindful Eating Questionnaire. Scores can range between 28 and 112, with higher scores indicating greater levels of mindful eating
Self-compassion | Baseline
  As measured by the Self-Compassion Scale Short Form. Scores range between 26 and 130, with higher scores indicating greater levels of self-compassion
Change in intuitive eating | Baseline, week 7, 24-week follow-up
  As measured by the Intuitive Eating Scale. Scores can range from 21 to 105, with higher scores indicating greater levels of intuitive eating
Cognitive restraint | Baseline
  As measured by the cognitive restraint subscale of the Three Factor Eating Questionnaire. Scores for this subscale range between 3 and 12, with higher scores indicating greater levels of cognitive restraint

CONTACTS AND LOCATIONS:
Overall Officials: Bärbel Knauper, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada